CLINICAL TRIAL: NCT00932503
Title: Do Triclosan Coated Sutures Reduce Wound Infections After Hepatobiliary Surgery? A Prospective Non Randomized Clinical Pathway Driven Study.
Brief Title: Antiseptic Sutures and Wound Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Principal Investigator, Christoph Justinger, Christoph Justinger, MDDepartment of General, Visceral, Vascular, and Pediatric Surgery, University Hospital, Saarland
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Vicryl plus 1
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Wound Infection
Keywords: Vicryl plus; wound infection; coated suture material; open abdominal surgery; transverse laparotomy
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PDS II (No Intervention): PDS II® loop suture was used for abdominal wall closure
- Vicryl plus (Active Comparator): antiseptic coated "Vicryl plus" was used for abdominal wall closure
  Interventions: Device: Vicryl plus

INTERVENTIONS:
Device: Vicryl plus — triclosan-coated polyglactin 910 suture materials with antiseptic activity (Vicryl plus®, Ethicon GmbH, Norderstedt, Germany)
  Other Names: Vicryl plus®
  Arms: Vicryl plus

SUMMARY:
The aim of this study was to ascertain if the use of Vicryl plus® reduced the number of wound infections after transverse laparotomy comparing to polydioxanon suture.

DETAILED DESCRIPTION:
All patients are treated using clinical pathways (CP) to standardise surgical procedures in our high volume centre. Part of the clinical process management was the standardisation of wound incision and abdominal wall closure.

Wound closure is achieved by a two-layer technique using continuous absorbable loop suture. The suture length to incision length ratio is at least 4:1. The running sutures are 1 cm apart and at least 1.5 cm from the wound edge 14. In the first timeperiod (TP1), the CP step for fascia closure foresees a PDS loop suture (PDS II®, 150 cm, Ethicon GmbH, Norderstedt, Germany). After the recruitment of 400 patients, that CP step is altered to the use of a triclosan-coated polyglactin 910 loop suture (Vicryl plus®, 150 cm, Ethicon GmbH, Norderstedt, Germany). The primary outcome is the number of wound infections. Patients demographic and disease as well as procedure related data are collected in a clinical information system (ISHmed on SAP platform, GSD, Berlin, Germany) prospectively. Risk factors for poor wound healing, such as operation time, patients age, sex, body mass index, blood loss, peritonitis, antibiotics, and performance level classified according to the American Society of Anesthesiologists (ASA), are collected prospectively to compare the two groups.

ELIGIBILITY:
Inclusion Criteria:

* surgical pathologies accessed via transverse abdominal incision
* primary fascial closure

Exclusion Criteria:

* pregnancy
* age under 18 years
* open abdominal treatment
* known hypersensitivity agains PDS/Vicryl/Triclosan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 839 (Actual)
Dates: Start 2003-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the number of wound infections. | 10 days after demission of patient from hospital

SECONDARY OUTCOMES:
The secondary outcome was the number of incisional hernia | follow up points: 6 month, 1 year, 2 years and 3 years
  long time follow up analyzing the number of incisional hernia after laparotomy comparing Vicryl plus and PDS II

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Justinger, M.D., Principal Investigator — Department of General, Visceral, Vascular and Pediatric Surgery, University of Saarland, D-66421 Homburg/Saar, Germany; Martin K Schilling, M.D., Study Director — Department of General, Visceral, Vascular and Pediatric Surgery, University of Saarland, D-66421 Homburg/Saar, Germany
Locations (1):
- Department of General, Visceral, Vascular and Pediatric Surgery, University of Saarland, D-66421 Homburg/Saar, Germany, Homburg/Saar, Germany

REFERENCES:
- [Result] Justinger C, Moussavian MR, Schlueter C, Kopp B, Kollmar O, Schilling MK. Antibacterial [corrected] coating of abdominal closure sutures and wound infection. Surgery. 2009 Mar;145(3):330-4. doi: 10.1016/j.surg.2008.11.007. Epub 2009 Jan 25. PMID 19231586